CLINICAL TRIAL: NCT00221104
Title: Secondary Prevention With HMG-CoA Reductase Inhibitor Against Stroke
Brief Title: Japan Statin Treatment Against Recurrent Stroke (J-STARS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government); Hiroshima University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: J-STARS; C000000207 (Other: UMIN CTR)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2017-06

CONDITIONS: Ischemic Stroke
Keywords: stroke; brain ischemia; cerebrovascular accident; statin; hydroxymethylglutaryl-CoA reductase inhibitors; cholesterol; hypercholesterolemia; hyperlipidemia; multicenter studies; prospective studies; endpoint determination; randomized controlled trials; recurrence; pravastatin
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Ischemia; Hypercholesterolemia; Hyperlipidemias; Recurrence | interventions — Pravastatin

ARMS (2):
- Pravastatin (Active Comparator): Patient has 10mg oral administration of Pravastatin per day. It starts within one month from their entry and continues every day until the end of the study or its endpoints.
  Interventions: Drug: Pravastatin
- No intervention (No Intervention): Patient has no intervention.

INTERVENTIONS:
Drug: Pravastatin
  Arms: Pravastatin

SUMMARY:
Although hyperlipidemia is not always the risk factor of stroke, inhibition of 3-hydroxy-3-methylglutaryl-coenzyme A(HMG-CoA) reductase can decrease the incidence of stroke in the patient with ischemic heart disease. The neuroprotective mechanism beyond cholesterol lowering should be expected to attenuate inflammation and atherosclerosis. The present study hypothesizes if pravastatin prevents recurrent stroke in the ischemic stroke patients with safety.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke except for cardiogenic embolism, from 1 month to 3 years after onset
* Hyperlipidemia and total cholesterol level of 180-240mg/dl without the prescription of statin within previous 30 days
* Able to visit outpatient department
* Informed consent on the form.

Exclusion Criteria:

* Ischemic stroke of other determined cause according to the TOAST classification
* Ischemic heart disease and necessary to use statin
* Hemorrhagic disorders
* Platelet count <=100,000/ul within 3 months prior to study start
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>= 100IU/L within 3 months prior to study start
* Serum creatinine >=2.0mg/dl within 3 months prior to study start
* A scheduled operation
* The presence of malignant disorder

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1578 (Actual)
Dates: Start 2004-03-01; Primary Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masayasu Matsumoto, MD, PhD, Principal Investigator — Hiroshima University Hospital
Locations (1):
- Hiroshima University, Hiroshima, Japan

REFERENCES:
- [Derived] Hosomi N, Kitagawa K, Nagai Y, Nakagawa Y, Aoki S, Nezu T, Kagimura T, Maruyama H, Origasa H, Minematsu K, Uchiyama S, Matsumoto M; J-STARS Collaborators. Desirable Low-Density Lipoprotein Cholesterol Levels for Preventing Stroke Recurrence: A Post Hoc Analysis of the J-STARS Study (Japan Statin Treatment Against Recurrent Stroke). Stroke. 2018 Apr;49(4):865-871. doi: 10.1161/STROKEAHA.117.018870. Epub 2018 Mar 6. PMID 29511130
- [Derived] Hosomi N, Nagai Y, Kitagawa K, Nakagawa Y, Aoki S, Nezu T, Kagimura T, Maruyama H, Origasa H, Minematsu K, Uchiyama S, Matsumoto M; J-STARS collaborators. Pravastatin Reduces the Risk of Atherothrombotic Stroke when Administered within Six Months of an Initial Stroke Event. J Atheroscler Thromb. 2018 Mar 1;25(3):262-268. doi: 10.5551/jat.40196. Epub 2017 Sep 16. PMID 28924103
- [Derived] Nakamura M, Fukukawa T, Kitagawa K, Nagai Y, Hosomi N, Minematsu K, Uchiyama S, Matsumoto M, Miyamoto Y; for J-STARS collaborators. Ten-year standardization of lipids and high-sensitivity C-reactive protein in a randomized controlled trial to assess the effects of statins on secondary stroke prevention: Japan Statin Treatment Against Recurrent Stroke. Ann Clin Biochem. 2018 Jan;55(1):128-135. doi: 10.1177/0004563217693651. Epub 2017 Jul 10. PMID 28135841
- See also: Japan Statin Treatment Against Recurrent Stroke (J-STARS) only in Japanese — http://jstars.umin.ne.jp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from March 2004 and February 2009 recruited at 123 clinical sites in Japan
Pre-assignment Details: Participants were randomly assigned to the pravastatin group or the control with 1:1 allocation rate. The patient allocation was dynamically balanced with the stroke subtype (atherothrombotic infarction vs. others), high blood pressure (≥150/90 mmHg vs. not), and diabetes mellitus (absence vs. presence) between the two groups.
Groups:
- Pravastatin Group: The administration was initiated within 1 month after randomization, and the treatment was continued until final observation. Diet and exercise therapies were reinforced when the total cholesterol levels consistently exceeded 6·21 mmol/L (240 mg/dL) at routine clinical visits. Increase of pravastatin dose or addition of other non-statin drugs (such as ion exchange resin, eicosapentaenoic acid and ezetimibe) was allowed only when such reinforcements were insufficient. Even under such conditions, use of other statins (such as simvastatin and atorvastatin) was prohibited.
- Control Group: The administration of any statin was prohibited, although use of other non-statin drugs was allowed when necessary.
Period: Overall Study
Arm/Group | Pravastatin Group | Control Group
Started | 793 | 785
Completed | 710 | 709
Not Completed | 83 | 76
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 42 | 29
Not completed — Others | 37 | 47

BASELINE CHARACTERISTICS:
Population: intention to treat
Groups:
- Pravastatin: The administration was initiated within 1 month after randomization, and the treatment was continued until final observation. Diet and exercise therapies were reinforced when the total cholesterol levels consistently exceeded 6·21 mmol/L (240 mg/dL) at routine clinical visits. Increase of pravastatin dose or addition of other non-statin drugs (such as ion exchange resin, eicosapentaenoic acid and ezetimibe) was allowed only when such reinforcements were insufficient. Even under such conditions, use of other statins (such as simvastatin and atorvastatin) was prohibited.
- Total: Total of all reporting groups
Arm/Group | Pravastatin | Control Group | Total
Number analyzed (Participants) | 793 | 785 | 1578
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 335 | 329 | 664
  >=65 years | 458 | 456 | 914
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 243 | 491
  Male | 545 | 542 | 1087
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 793 | 785 | 1578
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 793 | 785 | 1578
Ischemic stroke subtype [Number; unit: participants]
  Atherothrombotic infarction | 195 | 206 | 401
  Lacunar infarction | 502 | 504 | 1006
  Infarction of undetermined etiology | 96 | 75 | 171
High blood pressure [Number; unit: participants] — The high blood pressure was defined ≥150/90 mmHg at baseline.
  participants
    Yes | 308 | 309 | 617
    No | 485 | 476 | 961
Diabetes mellitus [Number; unit: participants]
  Yes | 185 | 184 | 369
  No | 608 | 601 | 1209

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Stroke and TIA
Description: Incidence rate of patients with recurrent stroke of any type or transient ischemic attack (TIA)
Time Frame: up to 5 years
Population: intention to treat
Measure: Number (95% Confidence Interval); unit: events /100 person-years
Arm/Group | Pravastatin | Control Group
Number analyzed (Participants) | 793 | 785
events /100 person-years | 2.56 [2.04 to 3.08] | 2.65 [2.12 to 3.18]
Statistical Analysis 1: Comparison: Pravastatin vs Control Group; the stratification factors at randomization: stroke subtype (atherothrombotic infarction vs. others), high blood pressure (≥150/90 mmHg vs. not), and diabetes mellitus (absence vs. presence); Test type: Superiority or Other; p = 0.8234, Stratified log-rank test; log-rank test adjusted for the stratification factors at randomization: stroke subtype, high blood pressure, and diabetes mellitus; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.73 to 1.29] — the adjusted hazard ratio (HR) and the 95% confidence interval (CI) were calculated by the Cox proportional hazard model with for the stratification factors at randomization: stroke subtype, high blood pressure, and diabetes mellitus

2. Secondary Outcome: Incidence Rate of Atherothrombotic Infarction
Description: Incidence rate of patients with atherothrombotic infarction
Time Frame: up to 5 years
Population: intention to treat
Measure: Number (95% Confidence Interval); unit: events /100 person-years
Arm/Group | Control Group | Pravastatin
Number analyzed (Participants) | 785 | 793
events /100 person-years | 0.65 [0.40 to 0.91] | 0.21 [0.06 to 0.35]
Statistical Analysis 1: Comparison: Control Group vs Pravastatin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0047, Stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.15 to 0.74] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Incidence Rate of Lacunar Infarction
Description: Incidence rate of patients with lacunar infarction
Time Frame: up to 5 years
Population: intention to treat
Measure: Number (95% Confidence Interval); unit: events /100 person years
Arm/Group | Pravastatin | Control Group
Number analyzed (Participants) | 793 | 785
events /100 person years | 1.26 [0.90 to 1.63] | 1.01 [0.69 to 1.33]
Statistical Analysis 1: Comparison: Pravastatin vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3075, Stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.81 to 1.91] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Incidence Rate of Cardioembolic Infarction
Description: Incidence rate of patients with cardioembolic infarction
Time Frame: up to 5 years
Population: intention to treat
Measure: Number (95% Confidence Interval); unit: events /100 person-years
Arm/Group | Pravastatin | Control Group
Number analyzed (Participants) | 793 | 785
events /100 person-years | 0.18 [0.05 to 0.32] | 0.08 [0.00 to 0.16]
Statistical Analysis 1: Comparison: Pravastatin vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1986, Stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 2.36, 95% CI 2-sided [0.61 to 9.14] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Incidence Rate of Intracranial Hemorrhage
Description: Incidence rate of patients with intracranial hemorrhage
Time Frame: up to 5 years
Population: intention to treat
Measure: Number (95% Confidence Interval); unit: events /100 person-years
Arm/Group | Pravastatin | Control Group
Number analyzed (Participants) | 793 | 785
events /100 person-years | 0.29 [0.12 to 0.46] | 0.31 [0.14 to 0.49]
Statistical Analysis 1: Comparison: Pravastatin vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9953, Stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.45 to 2.22] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Mean length of follow-up was 4.89 years.
Description: In the study AE form of clinical study CRF was not prepared. When serious adverse events (SAEs) in the study period were observed, SAEs were reported to principal investigator. AE/SAE were not observed at this study and those were spontanious reports from investigators. So the number at risk SAE (780) is not consistent with number participated (793). In regards to the Other AE, the meaning of number of participants at risk"0" here is because it were not monitored/ assessed.
Arm/Group | Pravastatin Group | Control Group
Serious Adverse Events (participants affected / at risk) | 188/780 | 164/785
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pravastatin Group (N=780) | Control Group (N=785)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 3 | 3
Angina unstable (Cardiac disorders) | 2 | 6
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 4
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Atrioventricular block second d (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 6 | 8
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 2
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 5 | 12
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2
Vertigo positional (Ear and labyrinth disorders) | 2 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 9 | 10
Cataract diabetic (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 4
Retinal artery occlusion (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal polyp (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 2 | 1
Colonic polyp (Gastrointestinal disorders) | 9 | 7
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diverticulitis intestinal haemo (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorr (Gastrointestinal disorders) | 2 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 2
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 3 | 5
Intestinal obstruction (Gastrointestinal disorders) | 2 | 3
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal haemorrh (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 2
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 43 | 35
Hernia (General disorders) | 1 | 0
Malaise (General disorders) | 4 | 0
Multi-organ failure (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 1
Swelling (General disorders) | 1 | 0
Therapy responder (General disorders) | 1 | 0
Disuse syndrome (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 2
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 3 | 1
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Hepatitis B (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 14 | 11
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 2
Pyothorax (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Encephalitis brain stem (Infections and infestations) | 1 | 0
Infected epidermal cyst (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 2
Biliary tract infection (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 6 | 4
Fracture (Injury, poisoning and procedural complications) | 12 | 10
Injury (Injury, poisoning and procedural complications) | 3 | 2
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Median nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Heat illness (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase in (Investigations) | 0 | 1
Catheterisation cardiac (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate co (Metabolism and nutrition disorders) | 8 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 6
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour of the duodenu (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 7
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Autonomic nervous system imbala (Nervous system disorders) | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 5 | 4
Cerebral haemorrhage (Nervous system disorders) | 11 | 9
Cerebral infarction (Nervous system disorders) | 17 | 19
Cerebrovascular accident (Nervous system disorders) | 0 | 3
Convulsion (Nervous system disorders) | 2 | 0
Dementia (Nervous system disorders) | 4 | 3
Dizziness (Nervous system disorders) | 4 | 4
Embolic stroke (Nervous system disorders) | 7 | 1
Epilepsy (Nervous system disorders) | 2 | 4
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 3
Loss of consciousness (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 2
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 1
Parkinsonism (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 7 | 9
Reversible ischaemic neurologic (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 43 | 39
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1
Spinal cord infarction (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 3
Cerebral artery stenosis (Nervous system disorders) | 1 | 2
Thrombotic cerebral infarction (Nervous system disorders) | 8 | 24
Dementia with Lewy bodies (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 3 | 3
Depression (Psychiatric disorders) | 2 | 0
Dissociative disorder (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 2 | 0
Nephritis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 2 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 3
Renal failure chronic (Renal and urinary disorders) | 1 | 2
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 2
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary d (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Social stay hospitalisation (Social circumstances) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Gastrostomy (Surgical and medical procedures) | 1 | 0
Coronary angioplasty (Surgical and medical procedures) | 1 | 1
Hepatectomy (Surgical and medical procedures) | 0 | 1
Removal of foreign body (Surgical and medical procedures) | 1 | 0
Laminaplasty (Surgical and medical procedures) | 1 | 0
Percutaneous coronary intervent (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 4 | 3
Aortic dissection (Vascular disorders) | 3 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Thrombophlebitis migrans (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Aortic rupture (Vascular disorders) | 1 | 0
Infarction (Vascular disorders) | 0 | 1
Artery dissection (Vascular disorders) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 1
Arteriosclerosis obliterans (Vascular disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No